CLINICAL TRIAL: NCT02464696
Title: A Prospective Randomized Controlled Trial of Early Non-Invasive Positive Pressure Ventilation in Patients With Hypoxemic Respiratory Failure and Malignancies
Brief Title: Non-invasive Ventilation in Reducing the Need for Intubation in Patients With Cancer and Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0165; NCI-2015-01514 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0165 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Methylprednisolone; exifone; Medrol Veriderm; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (NIPPV therapy) (Experimental): Patients undergo intermittent NIPPV, with the recommended schedule comprising 2 hours on NIPPV followed by =< 2 hours off NIPPV and continuous NIPPV at night or while sleeping for 8 hours per day, for 28 days or until discharged from the hospital.
  Interventions: Drug: Methylprednisolone; Device: Positive Air Pressure Device
- Arm B (high flow oxygen therapy) (Active Comparator): Patients continue to receive high flow nasal cannula oxygen therapy using current protocol for titration of high flow oxygen therapy for 28 days or until discharged from the hospital. Patients may receive NIPPV if they develop evidence of accessory muscle use with breathing or at the discretion of the treating physician.
  Interventions: Drug: Methylprednisolone; Procedure: Oxygen Therapy

INTERVENTIONS:
Drug: Methylprednisolone — IPS cohort only
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Procedure: Oxygen Therapy — Receive high flow oxygen therapy
  Other Names: supplemental oxygen therapy
  Arms: Arm B (high flow oxygen therapy)
Device: Positive Air Pressure Device — Undergo NIPPV
  Arms: Arm A (NIPPV therapy)

SUMMARY:
This randomized clinical trial studies how well non-invasive ventilation works in reducing the need for intubation, or placement of a tube in the windpipe, in patients with cancer and respiratory failure. Respiratory failure is a condition in which not enough oxygen passes from the lungs to the blood, and is a common cause of admission to the emergency room in patients with hematological and solid tumor patients. Non-invasive positive pressure ventilation (NIPPV) is a method of delivering oxygen using a mask. It is not yet known whether NIPPV is better at improving the amount of oxygen in the blood, reducing shortness of breath, and the need for intubation than standard high flow oxygen (a tube with 2 prongs placed in the nostrils) in patients with cancer and respiratory failure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the percent of patients who meet criteria for intubation within 28 days of study inclusion.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (NIPPV THERAPY): Patients undergo intermittent NIPPV, with the recommended schedule comprising 2 hours on NIPPV followed by =< 2 hours off NIPPV and continuous NIPPV at night or while sleeping for 8 hours per day, for 28 days or until discharged from the hospital.

ARM B (HIGH FLOW OXYGEN THERAPY): Patients continue to receive high flow nasal cannula oxygen therapy using current protocol for titration of high flow oxygen therapy for 28 days or until discharged from the hospital. Patients may receive NIPPV if they develop evidence of accessory muscle use with breathing or at the discretion of the treating physician.

IDIOPATHIC PULMONARY SYNDROME (IPS) SUBGROUP (INCLUDING DIFFUSE ALVEOLAR HEMORRHAGE): Patients with IPS receive methylprednisolone daily on days 0-48 and every other day (QOD) on days 49-55 in parallel with NIPPV or oxygen therapy, with a taper at the discretion of the treating physician.

After completion of study, patients are followed up until day 100.

ELIGIBILITY:
Inclusion Criteria:

* Partial pressure of arterial oxygen (PaO2):fraction of inspired oxygen (FiO2) ratio =< 300 mmHg OR a peripheral capillary oxygen saturation (SaO2):FiO2 =< 357
* Have a diagnosed malignancy
* Chest radiograph or computed tomography (CT) scan within =< 3 months prior to study enrollment rules out primary or metastatic malignancy in the lungs or pleural space as a significant cause of respiratory insufficiency
* Probability of survival is at least 6 months

Exclusion Criteria:

* Presence of do not resuscitate (DNR)/do not intubate (DNI) orders at study entry
* Clinical evidence of left heart failure as the main etiology for respiratory compromise
* Evidence of active intrathoracic malignancy (primary or metastatic) in the lungs or pleural space that is a significant cause of respiratory insufficiency
* Patients with acute chronic obstructive disease exacerbation as the primary etiology for respiratory failure
* Evidence of accessory respiratory muscle use with breathing
* Shock (need for vasopressor therapy or mean arterial pressure [MAP] < 60 despite fluid administration)
* Oliguric acute renal failure (urine output < 500 ml/day) unless already on hemodialysis
* Patient already on NIPPV at the time of screening
* pH < 7.30 or partial pressure of carbon dioxide (pCO2) > 50 (if available)
* Fixed upper airway obstruction
* Airway or facial trauma that would hinder the use of a NIPPV mask
* Uncontrolled tachy or bradyarrhythmia or active myocardial ischemia defined as either: atrial fibrillation with rapid ventricular response (heart rate [HR] > 120 beats per minute [bpm]), ventricular tachycardia or nonsustained ventricular tachycardia (any rate), supraventricular tachycardia (any rate), third degree heart block (any rate), heart rate less than 40 beats per minute (regardless of the rhythm)
* Active myocardial ischemia defined as a clinical presentation at the time of screening consistent with acute coronary syndrome which includes unstable angina and electrocardiogram (EKG) changes suggestive of an either an acute ST elevation myocardial infarction (new ST elevations or new left bundle branch block) or acute non-ST elevation myocardial infarction (new ST depressions, new T wave inversions)
* Glasgow Coma Scale (GCS) < 8 or inadequate airway protective reflexes
* Undrained pneumothorax/pneumomediastinum
* Copious secretions (> 20 cc's of sputum production per hour or significant hemoptysis defined as > 100 cc's of hemoptysis in a 24 hour period
* Risk for gastric aspiration (ie; ileus, esophageal or bowel obstruction, active vomiting)
* Recent esophageal, gastric or bowel surgery (within 3 weeks of study enrollment)
* Inability to cooperate with NIPPV
* Refusal to receive NIPPV
* Respiratory arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2015-10-06 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients who require intubation or meet criteria for intubation | Up to 28 days from study inclusion
  Fisher's exact test or a chi-squared test will be used to assess the association between two categorical variables. The intubation rate by 28 days and 95% confidence intervals will be estimated for each treatment arm. Logistic regression will be utilized to assess the effect of patient prognostic factors on the intubation rate by 28 days.

SECONDARY OUTCOMES:
Time to intubation | Up to 28 days
  The Kaplan-Meier method will be used to estimate the time-to-event distribution for each treatment group, and the median time will be provided. The log-rank test will be used to examine the time-to-event distribution of the active treatment group versus that of the control. Time to intubation rate at different time points will be provided by treatment group (i.e. at 7 days, 14 days, 21 days, and 28 days). Since there might be other competing risks for intubation, a competing risk analysis will be performed treating these early events as a competing event for intubation.
Intensive care unit length of stay | Up to 28 days
  Descriptive statistics, including the mean, standard deviation, median, and range, will be provided. The t-test or Wilcoxon's rank sum test will be used to evaluate the difference between the non-invasive positive pressure ventilation (NIPPV) arm and the control arm.
Hospital length of stay | Up to 28 days
  Descriptive statistics, including the mean, standard deviation, median, and range, will be provided. The t-test or Wilcoxon's rank sum test will be used to evaluate the difference between the NIPPV arm and the control arm.
Change in partial pressure of arterial oxygen (PaO2):fraction of inspired oxygen (FiO2) ratio | Baseline up to 28 days
  Descriptive statistics, including the mean, standard deviation, median, and range, will be provided. The t-test or Wilcoxon's rank sum test will be used to evaluate the difference between the NIPPV arm and the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Rathi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org